CLINICAL TRIAL: NCT00326196
Title: CSP #557 - Coronary Artery Revascularization in Diabetes (VA CARDS)
Brief Title: Coronary Artery Revascularization in Diabetes
Acronym: VA CARDS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participant enrollment
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 557
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Coronary Disease; Diabetes; PCI
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Diabetes Mellitus | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI (Active Comparator): Percutaneous coronary intervention
  Interventions: Device: Percutaneous coronary intervention (PCI); Procedure: Coronary artery bypass graft (CABG)
- CABG (Active Comparator): Coronary artery bypass graft (CABG)
  Interventions: Procedure: Coronary artery bypass graft (CABG)

INTERVENTIONS:
Device: Percutaneous coronary intervention (PCI) — percutaneous coronary stenting with drug eluding stents
  Arms: PCI
Procedure: Coronary artery bypass graft (CABG) — coronary bypass

SUMMARY:
This is a randomized, multi-site, clinical trial comparing percutaneous coronary stenting (PCI) with drug eluding stents to coronary bypass for angiographically significant coronary artery disease in diabetes. The hypothesis being tested is that a strategy of surgical revascularization is superior to percutaneous intervention in preventing death or myocardial infarction in diabetics with severe ischemic heart disease.

DETAILED DESCRIPTION:
Diabetic patients (HbA1c greater than 6.0% if treated or greater than 6.9% untreated) with severe ischemic heart disease and clinical indications for coronary revascularization will be screened and, if agreeable, entered into the study. Qualified patients unwilling to participate in the randomized trial will be approached for participation in a Registry that will collect computerized health data. The study consists of a 4-year accrual period. The median follow-up will be 3.7 years with a maximum of six years and a minimum of two years. Six sites will begin recruitment in the first year followed by nine additional sites for the remaining three years. The study is powered to detect a 40% relative difference between the groups in time to death or MI with a two-sided, type I error of 5% and a power of 90%.

ELIGIBILITY:
Inclusion Criteria:

Patients with diabetes with severe coronary artery disease General Inclusion Criteria

1. Age at least 18 years old
2. Patients with either Type I or Type II diabetes with a documented HbA1c greater than site ULN (If not on diabetic medication must be confirmed by a blood glucose of >126 mg/dL fasting, or >200mg/dL non-fasting); OR on diabetic medication with a documented physician diagnosis of diabetes mellitus.
3. No child bearing potential (if female)
4. Patient competent to provide consent

   Exclusion Criteria:

   General Exclusion Criteria
5. Congenital heart disease
6. Coronary bypass surgery within the preceding one year
7. Need for concomitant cardiac surgery
8. AHA Class III decompensated heart failure or AHA Class IV heart failure
9. Undergoing PCI for hemodynamic instability related to acute STEMI
10. History of a hemorrhagic stroke
11. Severe bleeding diathesis
12. History of chronic pancreatitis
13. A severe co-morbid condition that is expected to limit life to less than two years
14. Embolic stroke in the past six months
15. Significant GI bleed within the last one month
16. Lack of adequate surgical conduit
17. Sensitivity to clopidogrel (Plavix)
18. Sensitivity to glycoprotein IIb/IIIa inhibitors
19. Chronic systemic steroid use
20. Participation in another trial with active intervention
21. Patient unable to be adequately followed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2006-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoor Kamalesh, MD, Study Chair — Richard Roudebush VA Medical Center, Indianapolis
Locations (26):
- United States (26):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles HCS, Sepulveda, Sepulveda, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - VA Medical Center, Miami, Miami, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Asheville, Asheville, North Carolina
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Oklahoma City, Oklahoma City, Oklahoma
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Kamalesh M, Sharp TG, Tang XC, Shunk K, Ward HB, Walsh J, King S 3rd, Colling C, Moritz T, Stroupe K, Reda D; VA CARDS Investigators. Percutaneous coronary intervention versus coronary bypass surgery in United States veterans with diabetes. J Am Coll Cardiol. 2013 Feb 26;61(8):808-16. doi: 10.1016/j.jacc.2012.11.044. PMID 23428214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment occured at 23 VA medical centers and thestudy recruitment lasted from 8/25/2006 thru 3/24/2010.
Pre-assignment Details: Study participants were were pre-screened by Cath lab. The remaining participants were consented and screened for study eligibility.
Groups:
- Percutaneous Coronary Intervention: Initial revascularization with Percutaneous coronary intervention. Whenever possible, drug-eluting stents will be used in the percutaneous treatment. The use of multiple stents to achieve a "complete" revascularization will be encouraged in the PCI treatment
- Coronary Artery Bypass Graft: Initial revascularization with Coronary artery bypass graft (CABG). Multiple arterial conduits for suitable target vessels will be encouraged in the surgical treatment.
Period: Overall Study
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Started | 101 | 97
Completed | 101 | 97
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Percutaneous Coronary Intervention: Percutaneous coronary intervention
- Coronary Artery Bypass Graft: Coronary artery bypass graft (CABG)
- Total: Total of all reporting groups
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft | Total
Number analyzed (Participants) | 101 | 97 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (7.1) | 62.1 (7.4) | 62.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 100 | 96 | 196
Region of Enrollment [Number; unit: participants]
  United States | 101 | 97 | 198

OUTCOME MEASURES:

1. Primary Outcome: The Hypothesis Being Tested is That a Strategy of Initial Surgical Revascularization is Superior to Percutaneous Intervention in Preventing Death or Myocardial Infarction in Diabetics With Severe Ischemic Heart Disease Assessed up to 4 Years.
Description: Participants were monitored for up to 4 years. This is the number of particiapnts who have died or had at least one myocardial infarction.
Time Frame: Date of Death and non-fatal MI
Population: The number of participants for analysis was determined by intent to treat principal.
Measure: Number; unit: participants
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Number analyzed (Participants) | 101 | 97
participants | 21 | 16

ADVERSE EVENTS:
Time Frame: Date of Death and non-fatal MI, assessed up to 4 years.
Arm/Group | Percutaneous Coronary Intervention | Coronary Artery Bypass Graft
Serious Adverse Events (participants affected / at risk) | 23/101 | 46/97
Other Adverse Events (participants affected / at risk) | 7/101 | 67/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention (N=101) | Coronary Artery Bypass Graft (N=97)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (3)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 3 (3) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Thrombosis in device (General disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (3)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Coronary Intervention (N=101) | Coronary Artery Bypass Graft (N=97)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (6)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial disease (Cardiac disorders) | 0 (0) | 1 (1)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 0 (0) | 1 (1)
Incision site cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Graft complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 8 (8)
Pleuritic pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary oedema (Surgical and medical procedures) | 0 (0) | 1 (1)
Respiratory failure (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Transfusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Low participant recruitment led to the study being terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No